CLINICAL TRIAL: NCT06552806
Title: The Effect of a Multi-strain Probiotic SLAB51 (Sivomixx800®) on Acclimatization to High Altitude
Brief Title: The Effect of a Multi-strain Probiotic on Acclimatization to High Altitude
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Tatum Simonson, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 807971
Record Dates: First submitted 2023-07-06; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Probiotics

STUDY DESIGN:
Intervention Model Description: Repeated measurement double-blind, placebo controlled, cross-over study
Who Masked: Outcomes Assessor
Masking Description: Our collaborators Massimiliano Marazzato, PhD (Sapienza University of Rome) and Claudio de Simone, MD, PhD (https://www.probiotixx.info/en/about/) will provide both placebo and treatment samples codified, and their true formulation will be revealed to the investigators at UCSD after all the experiments and analysis are performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): SLAB51 will be administered orally each day during the four days at high altitude. Each dose of SLAB51 consists of one six-gram sachet dissolved in 100 mL of water, containing approximately 800 billion bacteria. Participants will receive, in one of their trips, one dose of SLAB51 after arrival to high altitude, then three times a day approximately every 5 hours upon waking during Days 2 and 3, and a final dose the morning of Day 4 of acclimatization.
  Interventions: Dietary Supplement: SLAB51
- Placebo group (Placebo Comparator): Placebo will be administered in the other trip, following the same schedule as SLAB51 as described above.
  Interventions: Dietary Supplement: SLAB51

INTERVENTIONS:
Dietary Supplement: SLAB51 — One dose of SLAB51 is administered after arrival to high altitude, then three times a day approximately every 5 hours upon waking during Days 2 and 3, and a final dose the morning of Day 4 of acclimatization.
  Other Names: Oxxyslab

SUMMARY:
The goal of this study is to learn if the probiotic SLAB51 (Sivomixx800®) works to enhance acclimatization to high altitude in humans. The main questions it aims to answer are:

Does SLAB51 improve oxygen saturation during high-altitude exposure? Researchers will compare SLAB51 to a placebo (a substance that contains no probiotic) to see if SLAB51 works to enhance high-altitude acclimatization.

Participants will:

Take SLAB51 or a placebo three times daily during two separate three-night acclimatization periods at high altitude, spaced at least six weeks apart.

Complete baseline measurements at sea level. Visit the high-altitude Barcroft Station (3,801 m) at the University of California White Mountain Research Center for physiological measurements and assessments.

Undergo assessments including oxygen saturation, ventilation, heart rate, blood pressure, sleep studies, cognitive assessments, exercise capacity, Acute Mountain Sickness scores, and provide blood, fecal, and urine samples for advanced analyses.

DETAILED DESCRIPTION:
Individuals will be recruited to participate in a double-blind, placebo controlled, cross-over study receiving placebo or the nutritional supplement probiotic SLAB51 (Sivomixx800®) during exposure to high altitude to test the effects of SLAB51 on high-altitude acclimatization.

Humans face significant physiological detriments when they ascend to high altitude due to hypobaric hypoxia, and physiological changes are crucial for acclimatization to this stressful environment. Currently, there are limited interventions to improve acclimatization to high altitude. The investigators conducting this study will test if the probiotic SLAB51 improves oxygen saturation and mitigates negative outcomes often experienced during acclimatization to high altitude through studies performed at sea level and at the high-altitude Barcroft Station (3,801 m) at the University of California White Mountain Research Center.

Preliminary studies indicate that ingestion of SLAB51 significantly improves oxygenation in humans during physical exercise in simulated altitude within a hypobaric chamber, in a pressurized airplane cabin during commercial flight, in premature born babies, and in COVID-19 patients. Here, the investigators explore whether ingestion of SLAB51 affects acclimatization to high altitude in healthy humans. Physiological measurements include oxygen saturation (O2 Sat or SpO2 during wakefulness and sleep, primary outcomes) as well as ventilation, heart rate, blood pressure, sleep studies, cognitive assessments, exercise capacity, measurement of the Acute Mountain Sickness score, and the collection of blood, fecal, and urine samples to further explored through transcriptomics, methylation, metabolomics, and proteomics. All measurements will be taken in up to 60 participants on two separate occasions separated by at least 6 weeks. Participants will complete all assessments, one baseline measurement obtained at sea level (0 - 300 m) and then twice during three-night acclimatization periods at Barcroft Station (3,801 m). At high altitude, participants will receive a treatment (placebo or SLAB51) upon arrival at Barcroft Station and then three times a day until departure from the high-altitude site. During the second portion of the study approximately six weeks later, participants will complete the same repeat assessments during a second three-night visit at Barcroft Station, where they will receive whichever treatment was not taken during the high-altitude exposure six weeks prior. Both participants and researchers performing the studies will be blinded to the treatment. Upon completion of the study, researchers will compare how participants acclimatized when they received SLAB51 versus when they received the placebo treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form. Participants must have the cognitive ability to consent to participate in this study.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Persons aged ≥ 18 years old or ≤ 65 years old.
* Women and men will be studied.
* We will recruit healthy participants, in good general health evidenced by medical history.
* Pregnancy test will be done previous to the beginning of the study. No other specific laboratory tests will be performed before the study.
* In the case of participants that can get pregnant, we ask them to use effective contraception at least 1 month previous to the beginning of the first trip, and in between the first and the second trip.
* Ability to take oral medication and be willing to adhere to the SLAB51 regimen.

Exclusion Criteria:

* No exclusion criteria based on languages spoken.
* No exclusion will be based on gender, race, socioeconomic status.
* History of cardiovascular or pulmonary disease, including HAPE and HACE.
* Female's menstrual phase and use of birth control pills will be documented, as hormones are reported to influence the control of breathing (Regensteiner et al. 1989). However, women under birth control will not be excluded from the study. Pregnant females will be excluded.
* Current smoker or tobacco use (more than 1 cigarette per day).
* Presence of systemic or local infection.
* Patients with history of chronic cardiac, pulmonary, renal, liver, neurological, or psychiatric disease (except controlled mood disorders), i.e., failure to achieve SaO2 > 95% when breathing supplemental oxygen (inspired PO2 = 200-225 mmHg, equivalent to 30% O2 at sea level).
* Cases of acute pancreatitis and acute hypersensitivity to gluten and lactose.
* Immunosuppressed patients.
* Participants with a BMI higher than 35.
* Participants will be asked to answer a survey (STOP-BANG Score for Obstructive Sleep Apnea, https://www.mdcalc.com/calc/3992/stop-bang-score-obstructive-sleep-apnea) to determine self-reported OSA. Patients with a STOP-Bang Score higher equal or higher than 3 will be excluded.
* Use of any medications or agents that might interfere with the physiological measurements, such as ventilation and heart rate, will result in exclusion from our study, such as ibuprofen, anti-hypertensives, benzodiazepines, sleep aids including melatonin, opioids, other narcotics/sedatives and acetazolamide.
* Participants must not have traveled above 2,500 m (8,202 feet) of elevation for 4 weeks prior to the initial baseline measurement at sea level and throughout the duration of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Oxygen saturation | At sea level (one day, one night) and all four days and three nights of the study at high altitude
  The effects of treatment group (probiotic or placebo) and timepoint on daytime SpO2 and mean nocturnal SpO2 will be determined by two-way analysis of variance (ANOVA) with a Bonferroni post hoc test.

SECONDARY OUTCOMES:
Hypoxic ventilatory response | At sea level (one day) and one day at high altitude
  Changes in ventilation due to the decrease of oxygen saturation (10%) and/or increase in carbon dioxide (5mmHg)
Heart rate | At sea level (one day, one night) and all four days at high altitude
  Heart rate measurement
Heart rate variability | At sea level (one day, one night) and all four days at high altitude
  Values of high frequency-low frequency ratio (HF/LF) of volunteers administered with SLAB51
Blood pressure | At sea level (one day, one night) and all four days at high altitude
  Blood pressure measurement
Sleep oxygen saturation | At sea level (one night) and all three nights of the study at high altitude
  Oxygen levels during sleep
Sleep apnea hypopnea index | At sea level (one night) and all three nights of the study at high altitude
  Number of times breathing stops and leads to a decrease of 3% oxygen saturation
Sleep oxygen desaturation index | At sea level (one night) and all three nights of the study at high altitude
  How often and how much a person's blood oxygen saturation drops (at least 4%) during sleep
Sleep duration | At sea level (one night) and all three nights of the study at high altitude
  How many hours and minutes a person sleeps during the night
Cancellation Pictures cognitive test | Two consecutive days at sea level, each of the four days at high altitude, and another time at sea level 1-2 weeks after returning from high altitude.
  A timed, tablet-based test of selective attention and inhibitory control
Contrast Sensitivity cognitive test | Two consecutive days at sea level, each of the four days at high altitude, and another time at sea level 1-2 weeks after returning from high altitude.
  Measures the ability to distinguish between fine increments of light and dark (contrast)
Digits-in-Noise cognitive test | Two consecutive days at sea level, each of the four days at high altitude, and another time at sea level 1-2 weeks after returning from high altitude.
  Presents trials of three sequential spoken digits against a broad-band, speech-shaped masker. The outcome measure is the threshold noise tolerance.
Spatial Release from Masking cognitive test | Two consecutive days at sea level, each of the four days at high altitude, and another time at sea level 1-2 weeks after returning from high altitude.
  Tests the ability to distinguish speech from competing speech using headphones and virtual spatial locations.
Trail Making cognitive test | Two consecutive days at sea level, each of the four days at high altitude, and another time at sea level 1-2 weeks after returning from high altitude.
  A measure of visual attention and task switching ability with outcome measures of response time and accuracy.
Oxygen saturation in submaximal exercise | At sea level (one day) and one day at high altitude
  Measurement of oxygen saturation during the final 30 seconds of submaximal exercise on a stationary bike
Lactate following submaximal exercise | At sea level (one day) and one day at high altitude
  Measurements of lactate following submaximal exercise on a stationary bike
Acute Mountain Sickness Score | At sea level (one day) and all four days of the study at high altitude
  Questionnaire to gauge how a person feels at high altitude. It defines AMS as the presence of headaches in addition to three other symptoms, including gastrointestinal symptoms, fatigue/weakness, and dizziness/lightheadedness. Each symptom is appointed a point on a scale from 0 to 3, with 0 being no effect and 3 being severe. A total score of 3 or greater, with the presence of headaches, in a setting of rapid ascent to high altitude, is diagnosed as acute mountain sickness.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - White Mountain Research Station, Bishop, California
  - University of California, San Diego, La Jolla, California

IPD SHARING:
Plan to Share IPD: No
Although general information of mean and standard error data will be indicated in the graphs used for this project, individual data will be shown in as dots in the exposed graphs, and in tables when this is not possible.